CLINICAL TRIAL: NCT00033904
Title: A Multi-Center, Randomized Phase III Study of Adjuvant Oncophage® Versus Observation in Subjects With High Risk of Recurrence After Surgical Treatment for Renal Cell Carcinoma
Brief Title: Survival Study Of Oncophage® vs. Observation In Patients With Kidney Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-100-12 Part I
Record Dates: First submitted 2002-04-12; First posted 2002-04-15 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Renal Cell Carcinoma
Keywords: Kidney Cancer, renal, immunotherapy, tumor,
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Neoplasms

INTERVENTIONS:
Drug: autologous human tumor-derived HSPPC-96

SUMMARY:
Determine whether patients receiving adjuvant HSPPC-96 treatment after surgically resected, locally advanced renal cell carcinoma have improved recurrence-free survival as compared to subjects with no adjuvant treatment.

DETAILED DESCRIPTION:
Primary Objective:

* The primary objective of this study is to determine whether subjects randomized to receive adjuvant HSPPC-96 after surgical resection of locally advanced renal cell carcinoma at high risk of recurrence, have improved recurrence-free survival as compared to subjects with no adjuvant treatment.

Secondary Objective:

* Determine whether subjects randomized to receive HSPPC-96 have improved survival as compared to subjects with no adjuvant treatment.
* Further characterize the safety profile of HSPPC-96.

ELIGIBILITY:
Pre-Surgery Inclusion Criteria:

* Primary-intact resectable renal cell cancer, without known distant metastasis and be scheduled to have surgery with curative intent;
* Tumor size greater than or equal to 5 cm OR macroscopic nodes OR renal vein thrombus OR vena cava thrombus by radiologic evaluation
* Performance status (Zubrod / ECOG-WHO scale)less than or equal to 1 and life expectancy of greater than three months, within 2 weeks of surgery.
* Women of child-bearing potential must have a negative urine or serum pregnancy test within 2 weeks of surgery.
* Signed written informed consent.

Pre-Surgery Exclusion Criteria:

* Prior chemo-, hormonal, immuno- or radiotherapy for renal cell cancer;
* History of primary or secondary immunodeficiency, or patients using immunosuppressive drugs, e.g. systemic corticosteroids, cyclosporin A;
* Current malignancies at other sites or previous other cancer within the last 5 years, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri or basal or squamous cell carcinoma of the skin;
* Embolization of the renal artery prior to nephrectomy;
* Known distant metastases;
* Active, uncontrolled infection or other serious medical illnesses.

Eligibility Assessment:

(between 2 weeks pre- and 4 weeks post-surgery)

Prior to randomization and entry into the tumor evaluation phase, all subjects must undergo testing to confirm that they are free of distant metastatic disease, and that they meet all other criteria.

Eligibility Criteria which must be assessed and confirmed prior to randomization:

* No evidence of metastatic or residual renal carcinoma as documented by all of the following: abdominal/pelvis CT scan; chest CT scan; and brain CT or MRI scan.
* Provide Antigenics with greater than or equal to 7 grams of viable tumor tissue
* Adequate bone marrow function.
* Adequate renal and hepatic function.
* Adequate cardiac function.
* Signed written informed consent.
* Patients must be willing to be followed during the course of tumor evaluation and follow-up phases.
* Male or female patients of child producing potential must agree to use adequate contraception during the treatment/observation phase of the study.
* Patients must not use any other investigational drug for four weeks prior to the start of the tumor evaluation phase and throughout the tumor evaluation phase of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650
Dates: Start 2000-06; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (76):
- United States (39):
  - Anchorage, Alaska
  - Tucson, Arizona
  - Los Angeles, California
  - San Francisco, California
  - Denver, Colorado
  - Farmington, Connecticut
  - Boca Raton, Florida
  - Miami, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Maywood, Illinois
  - Iowa City, Iowa
  - Kansas City, Kansas
  - Gretna, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Rochester, Minnesota
  - St Louis, Missouri
  - Albuquerque, New Mexico
  - Manhasset, New York
  - New York, New York
  - Rochester, New York
  - Charlotte, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Eugene, Oregon
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Fort Worth, Texas
  - Houston, Texas
  - South Burlington, Vermont
  - Richmond, Virginia
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Vienna, Austria
- Belgium (2):
  - Kortrijk
  - Liège
- Canada (7):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- France (4):
  - Lille
  - Strasbourg
  - Toulouse
  - Villejuif
- Israel (5):
  - Beer-Yaacob, Zerifin
  - Haifa
  - Holon
  - Jerusalem
  - Tel Litwinsky
- Norway (2):
  - Oslo
  - Stavanger
- Poland (7):
  - Bialystok
  - Gdansk
  - Kielce
  - Krakow
  - Lublin
  - Szczecin
  - Warsaw
- Spain (3):
  - Barcelona
  - Madrid
  - Valencia
- Sweden (4):
  - Gothenburg
  - Lund
  - Umeå
  - Uppsala
- United Kingdom (2):
  - Bristol
  - London

REFERENCES:
- [Derived] Wood C, Srivastava P, Bukowski R, Lacombe L, Gorelov AI, Gorelov S, Mulders P, Zielinski H, Hoos A, Teofilovici F, Isakov L, Flanigan R, Figlin R, Gupta R, Escudier B; C-100-12 RCC Study Group. An adjuvant autologous therapeutic vaccine (HSPPC-96; vitespen) versus observation alone for patients at high risk of recurrence after nephrectomy for renal cell carcinoma: a multicentre, open-label, randomised phase III trial. Lancet. 2008 Jul 12;372(9633):145-154. doi: 10.1016/S0140-6736(08)60697-2. Epub 2008 Jul 3. PMID 18602688